CLINICAL TRIAL: NCT01020604
Title: PROstaTE Cancer Treatment and Obesity in Zoladex-Astrazeneca Treated Patients Assessment of the Correlation Between Body Mass Index and Recurrence Among Zoladex Treated Prostate Cancer Patients
Brief Title: PROstaTE Cancer Treatment and Obesity in Zoladex-Astrazeneca Treated Patients
Acronym: PROTECT-Z
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OHU-ZOL-2009/1
Record Dates: First submitted 2009-11-20; First posted 2009-11-25 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Prostate Cancer; Obesity
Keywords: BMI; Prostate cancer; Recurrence
MeSH Terms: conditions — Prostatic Neoplasms; Obesity; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The reports on relationship of obesity and biochemical or clinical recurrence of prostate cancer are controversial. Several reports have shown that obesity is associated with increased risk of biochemical or clinical failure after radical prostatectomy. Other prospective studies have shown no adverse effect of obesity on long-term outcomes after prostatectomy. Limited reports are available on the impact of obesity on prostate cancer progression after radiotherapy. Primary: to assess percentage recurrence rate among normal weight and overweight or obese prostate cancer patients treated by adjuvant Zoladex therapy. Secondary: to determine the Quality of Life differences among normal and overweight or obese prostate cancer patients by a Quality of Life questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven prostate cancer patients being on adjuvant Zoladex treatment after primary therapy or on adjuvant therapy without primary curative therapy

Exclusion Criteria:

-Prostate cancer patients refractory to hormonal therapy, not agreeing to participate, allergy against treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult men treated by adjuvant goserelin therapy for at least 1 month after primary (curative) therapy of histologically proven, prostate cancer
Sampling Method: Probability Sample
Enrollment: 1376 (Actual)
Dates: Start 2009-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Percentage recurrence rate among normal weight and overweight or obese prostate cancer patients treated by adjuvant Zoladex therapy. | Every 3 months

SECONDARY OUTCOMES:
Quality of Life differences among normal and overweight or obese prostate cancer patients by a Quality of Life questionnaire | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Istvan Buzogany, Principal Investigator — Budapest City's Local Government "Péterfy Sándor" Hospital and Ambulatory Clinic
Locations (34):
- Hungary (34):
  - Research Site, Baja
  - Research Site, Barcs
  - Research Site, Békés
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Csongrád
  - Research Site, Debrecen
  - Research Site, Dunaharaszti
  - Research Site, Dunaújváros
  - Research Site, Győr
  - Research Site, Gyula
  - Research Site, Helvécia
  - Research Site, Jászberény
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Kiskunhalas
  - Research Site, Kőszárhegy
  - Research Site, Makó
  - Research Site, Miskolc
  - Research Site, Nagyvenyim
  - Research Site, Nyíregyháza
  - Research Site, Nyírpazony
  - Research Site, Orosháza
  - Research Site, Pápa
  - Research Site, Pécs
  - Research Site, Salgótarján
  - Research Site, Szeged
  - Research Site, Szekszárd
  - Research Site, Szentendre
  - Research Site, Székesfehérvár
  - Research Site, Szolnok
  - Research Site, Szombathely
  - Research Site, Tiszaföldvár
  - Research Site, Veszprém